CLINICAL TRIAL: NCT05669235
Title: Differences Between Women Who Have Suffered COVID-19 With Respect to Those Who Have Suffered Long Covid: Observational Study
Brief Title: Differences Between Women With COVID-19 and Long Covid
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, University of Valencia
Other Study IDs: OBS_LCOVID
Record Dates: First submitted 2022-12-29; First posted 2022-12-30 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: COVID-19; Long covid; Women
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long covid: Women who present symptoms after suffering from COVID-19, consistent with long covid.
  Interventions: Diagnostic Test: Questionnaires
- Covid: Women who have passed COVID-19 without consequences.
  Interventions: Diagnostic Test: Questionnaires

INTERVENTIONS:
Diagnostic Test: Questionnaires — A series of questionnaires will be carried out that assess both respiratory problems, depression and strength.

SUMMARY:
The coronavirus disease of 2019 (COVID-19) has infected more than 630 million people and resulted in more than 6.5 million deaths worldwide. Among the possible sequelae of the virus, a disorder called long COVID has shown to affect about 10% of those infected, mostly adult women, without comorbidities.

Long COVID corresponds to a multisystemic syndrome following the acute period of the disease, in which the person maintains persistent symptoms such as fatigue, dyspnea, cough, memory loss, muscle and joint pain, among others.

Now that time has passed, it is necessary to verify why there are women who present symptoms of long covid and others do not.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 65 years
* That they have passed COVID-19 at least once.
* Whether or not they have symptoms secondary to COVID-19.

Exclusion Criteria:

* They do not want to sign the informed consent.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women who have suffered from COVID-19 who have or have not had symptoms since then.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | Baseline
  Scale that measures fatigue, made up of 10 items rated from 1 to 5: 1. Never 2. Sometimes (think of a frequency of once a month or less, for example) 3. Regularly (for example, a couple of times a month) 4. often (think for example every week) 5. always (every day)

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale | Baseline
  The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases.
  Describes baseline dyspnea, but does not accurately quantify response to treatment of chronic obstructive pulmonary disease (COPD).
  Demonstrates at least moderate positive correlation with other dyspnea scores, including the baseline dyspnea index (BDI) and oxygen cost diagram (OCD). It measures the degree of dyspnea in 5 levels (from 0 to 4).
Quality of life (EQ-5D) | Baseline
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome.
Perceived Stress Scale (PSS) | Baseline
  A more precise measure of personal stress can be determined by using a variety of instruments that have been designed to help measure individual stress levels. The first of these is called the Perceived Stress Scale. The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The tool, while originally developed in 1983, remains a popular choice for helping us understand how different situations affect our feelings and our perceived stress. The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certain way. Although some of the questions are similar, there are differences between them and you should treat each one as a separate question. The best approach is to answer fairly quickly. That is, don't try to count up the number of times you felt a particular way; rather indicate the alternative that seems like a reasonable estimate.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The Patient Health Questionnaire 9-item depression scale (PHQ-9) and 7-item Generalized Anxiety Disorder scale (GAD-7) are among the best validated and most commonly used depression and anxiety measures, respectively.20-25 They have been used in hundreds of research studies, incorporated into numerous clinical practice guidelines, and adopted by a variety of medical and mental health care practice settings. Importantly, the PHQ-9 and GAD-7 are public domain measures available in more than 80 translations, many of which can be freely downloaded at www.phqscreeners.com. This paper uses data from 3 clinical trials to examine the reliability and convergent, construct, and factor structure validity as well as sensitivity to change of the Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) - a 16-item scale comprising the PHQ-9 and GAD-7 - as a composite measure of depression and anxiety.
Inventario de Depresión de Beck (BDI-2) | Baseline
  This test consists of 21 multiple-choice questions, where the subject in question who takes the test must assess on a scale of 0 to 3 the degree to which he personally identifies with the answer he has answered in it (where 0 is that you do not identify at all, being able to conclude that you do not present the symptoms on which the question is concerned; and 3 is that there is an absolute identification, for which, the subject would suffer from the symptoms). It is a test that is easy to perform, in which the subject would not spend more than 10 or 15 minutes doing it.
30 second sit-to-stand | Baseline
  Test that measures the number of times you can get up and sit down in a chair in 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No